CLINICAL TRIAL: NCT03730233
Title: Hiatal Hernia Repair by Tension-free Mesh Closure or Simple Suturing of the Diaphragmatic Hiatus. A Randomized, Double Blind Study With a 3-year Follow up.
Brief Title: Hiatal Hernia Repair by Tension-free Mesh Closure or Simple Suturing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/37-31/4
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Hiatal Hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: repair by tension-free mesh closure or simple suturing of the diaphragmatic
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomization process was initiated after general anesthesia had been induced and the group affiliation was determined by opening of a sealed envelope specifying the group assignment. The subsequent operation report, with information on the specific type of repair performed, was not included in the digital patient-chart. Instead, a hard copy was printed and kept in a sealed envelope, which was filed in a locked archive to maintain the patient, staff and clinical assessors blinded to the study group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tension-free (Active Comparator): Hiatal hernia repair by tension-free mesh closure
  Interventions: Procedure: Hiatal hernia repair by tension-free mesh closure
- Suturing (Active Comparator): Hiatal hernia repair by simple suturing of the diaphragmatic
  Interventions: Procedure: Hiatal hernia repair by simple suturing

INTERVENTIONS:
Procedure: Hiatal hernia repair by tension-free mesh closure
  Arms: Tension-free
Procedure: Hiatal hernia repair by simple suturing
  Arms: Suturing

SUMMARY:
One-hundred and fifty-nine patients undergoing Nissen fundoplication for symptomatic gastro-oesophageal reflux disease (GORD), who had a concomitant hiatal hernia of > 2 cm axial length, were randomized to closure of the diaphragmatic hiatus with either crural sutures alone or tension-free closure with a non-absorbable mesh. Primary outcome variable was the incidence of radiologically verified recurrent hiatal hernia. Secondary outcomes were per-and postoperative complications and courses, symptomatic recurrence rate, use of PPI, postoperative oesophageal acid exposure and Quality of Life.

DETAILED DESCRIPTION:
The basic principles behind successful surgical repair of the anatomy and function of the gastro-oesophageal junction (GOJ) in gastro-oesophageal reflux disease (GORD) is not only to encircle the distal oesophagus and GOJ by the fundic wrap but also to complete a transhiatal reduction of a concomitant hiatal hernia (type I, HH), aiming for a 2 - 3 cm intra-abdominal length of the of oesophagus and to transact a tension-free hiatal closure. The physiological and morphological characteristics of the diaphragmatic hiatus, however, carry a challenge for the selection of the ideal technique for surgical repair. The diaphragmatic hiatus consists of a three-dimensional structure in constant motion, which creates a border between the counteracting pressures prevailing in the abdominal and chest cavities, respectively. Following hernia reduction, the structural quality of the diaphragmatic pillars is usually weak, offering poor support for the subsequent closure with risk for high recurrence rates. These and other considerations have encouraged the exploration of mesh reinforcement to enhance the durability of the hiatal closure.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective laparoscopic total fundoplication
* symptomatic gastro oesophageal reflux disease (GORD) and HH of > 2 cm in axial length
* total esophageal acid exposure for more than 4 % of monitored time

Exclusion Criteria:

* if insufficient capacity prevailed to understand the study protocol,
* if the patient had undergone previous major upper gastrointestinal surgery (except for GORD or HH)
* ASA classification of >2 .

Ages: 20 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-01-11 (Actual); Primary Completion 2010-05-10 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Recurrent hiatal hernia | 12 month
  The incidence of radiologically verified recurrent hiatal hernia. Examined in the erect position after a 4-hour fast when 250 ml of low-density barium sulphate suspension (45% weight per volume) was ingested. The patients were instructed to drink the served volume within 30 seconds. Thereafter three sagittal spot films (35 x 35 cm) of the distal esophagus and GEJ were exposed 1, 2 and 5 minutes after the start of the barium ingestion (16). In

SECONDARY OUTCOMES:
Complications | from operation day up to 12 month
  Number of patients who had a bleeding or a leakage that requires a intervention, either blood transfusion or reoperation.
Proton pump inhibitor (PPI) | 12 month
  Use of PPI
Quality of Life, physical and mental score: SF-36 | 12 month
  The Swedish version of the validated global Short Form -36 (SF-36) questionnaire was used and data are presented as physical and mental summary component scores (PCS and MCS, respectively).
Postoperative oesophageal acid exposure | 12 month
  Ambulatory 24-hour pH-monitoring was performed by use of a slim-line dual probe catheter system (single-use, 2 sensors, 15 cm spacing, ø 1.8 mm, Medtronic A/S, Skovlunde, Denmark). The oesophageal pH probe was positioned 5 cm above the upper border of the LOS as determined by manometry. Total time in percent of the total recording time with pH <4 was determined
Gastrointestinal symptom rating scale (GSRS) | 12 month
  A validated questionnaire containing five dimensions of abdominal symptoms (gastroesophageal reflux, abdominal pain, indigestion, obstipation and diarrhea).
Dysphagia | 12 month
  Dysphagia for liquids and solids were recorded within a four-graded scale stating the frequency of dysphagia episodes with an arbitrary (empirical) cut off for clinical significance. The same dysphagia scoring was also used in a previous rct, from the same institution, comparing different types of antireflux procedures in open surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Professor, Principal Investigator — Karolinska Institutet

REFERENCES:
- [Derived] Analatos A, Hakanson BS, Lundell L, Lindblad M, Thorell A. Tension-free mesh versus suture-alone cruroplasty in antireflux surgery: a randomized, double-blind clinical trial. Br J Surg. 2020 Dec;107(13):1731-1740. doi: 10.1002/bjs.11917. Epub 2020 Sep 16. PMID 32936951